CLINICAL TRIAL: NCT06260722
Title: A Phase 3, Randomized, Multicenter, Open-label Study to Investigate the Efficacy and Safety of Retatrutide Once Weekly Compared With Semaglutide Once Weekly in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Metformin With or Without SGLT2 Inhibitor (TRANSCEND-T2D-2)
Brief Title: Effect of Retatrutide Compared With Semaglutide in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Metformin With or Without SGLT2 Inhibitor (TRANSCEND-T2D-2)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18805; J1I-MC-GZBZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Incretins
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases | interventions — retatrutide; semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Retatrutide Dose Level 1 (Experimental): Participants will receive retatrutide administered subcutaneously (SC).
  Interventions: Drug: Retatrutide
- Retatrutide Dose Level 2 (Experimental): Participants will receive retatrutide administered SC.
  Interventions: Drug: Retatrutide
- Semaglutide (Active Comparator): Participants will receive semaglutide administered SC.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Retatrutide — Administered SC.
  Other Names: LY3437943
  Arms: Retatrutide Dose Level 1; Retatrutide Dose Level 2
Drug: Semaglutide — Administered SC.
  Arms: Semaglutide

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of retatrutide compared with semaglutide in participants with Type 2 Diabetes and inadequate glycemic control with metformin with or without sodium-glucose cotransporter-2 inhibitor (SGLT2i). The study will last about 26 months and may include up to 24 visits.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes (T2D)
* Have HbA1c ≥ 7.0% (53 millimoles per mole (mmol/mol)) to ≤ 10.5% (91 mmol/mol)
* Have been on a stable diabetes treatment consisting of metformin ≥ 1500 milligrams per day (mg/day) with or without SGLT2i during 90 days prior to screening
* Are of stable weight for at least 90 days prior to screening
* Have a Body Mass Index (BMI) ≥ 25.0 kilograms per meter squared (kg/m^2)

Exclusion Criteria:

* Have Type 1 Diabetes (T1D)
* Have a history of ketoacidosis or hyperosmolar state or coma within the last 6 months prior to screening
* Have a history of severe hypoglycemia or hypoglycemia unawareness within the last 6 months prior to screening
* Are currently receiving or planning to receive treatment for diabetic retinopathy and/or macular edema
* Have an estimated glomerular filtration rate (eGFR) <45 milliliters/minute/1.73 meter squared (mL/min/1.73 m^2) or lower than the country-specific threshold for discontinuing metformin therapy per local label as determined by the central laboratory
* Have a prior or planned surgical treatment for obesity
* Have New York Heart Association Functional Classification IV congestive heart failure
* Have had an acute myocardial infarction, stroke, or were hospitalized for congestive heart failure within 90 days prior to screening
* Have a known clinically significant gastric emptying abnormality
* Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy for less than 5 years
* Have any lifetime history of a suicide attempt
* Had chronic or acute pancreatitis
* Have a family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia (MEN) syndrome Type 2
* Have taken prescribed or over-the-counter medication, or alternative remedies, intended to promote body weight reduction within 90 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hemoglobin A1c (HbA1c) (%) | Baseline, Week 80

SECONDARY OUTCOMES:
Change from Baseline in HbA1c (%) | Baseline, Week 80
Percentage of Participants Who Achieve HbA1c ≤ 6.5% | Week 80
Percentage of Participants Who Achieve HbA1c < 5.7% | Week 80
Percent Change from Baseline in Body Weight | Week 80
Change from Baseline in Body Weight | Baseline, Week 80
Percentage of Participants Who Achieve Weight Reduction of ≥ 5% | Week 80
Percentage of Participants Who Achieve Weight Reduction of ≥ 10% | Week 80
Percentage of Participants Who Achieve Weight Reduction of ≥ 15% | Week 80
Percentage of Participants Who Achieve HbA1c ≤ 6.5% and ≥ 10% Weight Reduction | Week 80
Percent Change from Baseline in Triglycerides | Week 80
Percent Change from Baseline in Non- high-density lipoprotein (HDL) Cholesterol | Week 80
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 80

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (77):
- United States (38):
  - University of Alabama - Department of Nutrition Sciences, Birmingham, Alabama
  - Neighborhood Healthcare Institute of Health, Escondido, California
  - Long Beach Research Institute, Long Beach, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Rancho Cucamonga Clinical Research, Rancho Cucamonga, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Arrow Clinical Trials, Daytona Beach, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - South Broward Research, Miramar, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Herman Clinical Research, Suwanee, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Pacific Diabetes & Endocrine Center, Honolulu, Hawaii
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Deaconess Clinic - Gateway Health Center, Newburgh, Indiana
  - IMA Clinical Research Monroe - Armand, Monroe, Louisiana
  - MedStar Health Research Institute (MedStar Physician Based Research Network), Hyattsville, Maryland
  - Brigham and Women's Hospital Diabetes Program, Boston, Massachusetts
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - Palm Research Center Sunset, Las Vegas, Nevada
  - NYC Research INC, Long Island City, New York
  - Medication Management, Greensboro, North Carolina
  - Remington Davis Clinical Research, Columbus, Ohio
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Central States Research, Tulsa, Oklahoma
  - The Corvallis Clinic, P.C., Corvallis, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Valley Institute of Research - Fort Worth, Fort Worth, Texas
  - Juno Research, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Medrasa Clinical Research, Wylie, Texas
  - Central Washington Health Services Association d/b/a Confluence Health, Wenatchee, Washington
  - IMA Clinical Research West Virginia, Morgantown, West Virginia
- Argentina (15):
  - CARE - Centro de Alergia y Enfermedades Respiratorias, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Stat Research S.A., Buenos Aires, Buenos Aires F.D.
  - CIPREC, Buenos Aires, Buenos Aires F.D.
  - Centro Médico Viamonte, Buenos Aires, Buenos Aires F.D.
  - Mautalen Salud e Investigación, Buenos Aires, Buenos Aires F.D.
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires, Buenos Aires F.D.
  - CEMEDIAB, C.a.b.a., Buenos Aires F.D.
  - Instituto Centenario, CABA, Buenos Aires F.D.
  - Centro Medico Privado San Vicente Diabetes, Córdoba, Córdoba Province
  - CIPADI - Centro Integral de Prevencion y Atencion en Diabetes, Godoy Cruz, Mendoza Province
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria, Santa Fe Province
  - Instituto de Investigaciones Clinicas Rosario, Rosario, Santa Fe Province
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Centro Diabetológico Dr. Waitman, Córdoba
- Canada (12):
  - University of Calgary - Clinical Trials Unit, Calgary, Alberta
  - Alberta Diabetes Institute, Edmonton, Alberta
  - Centricity Research Brampton Endocrinology, Brampton, Ontario
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Winterberry Research Inc., Hamilton, Ontario
  - The Wharton Medical Clinic Clinical Trials Inc, Hamilton, Ontario
  - Hamilton Medical Research Group, Hamilton, Ontario
  - Bluewater Clinical Research Group Inc., Sarnia, Ontario
  - Prime Health Clinical Research, Toronto, Ontario
  - Maple Leaf Research, Toronto, Ontario
  - Private Practice - Dr. Nigel Jagan, Whitby, Ontario
  - 9109-0126 Quebec Inc., Montreal, Quebec
- Mexico (10):
  - Diseno y Planeacion en Investigacion Medica, Guadalajara, Jalisco
  - RM Pharma Specialists, Mexico City, Mexico City
  - Hospital de Jésus, I.A.P., Mexico City, Mexico City
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, Mexico City, Mexico City
  - Instituto de Diabetes, Obesidad y Nutricion, Cuernavaca, Morelos
  - Cardiolink Clin Trials, Monterrey, Nuevo León
  - Clínica García Flores SC, Monterrey, Nuevo León
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Enclifar Ensayos Clínicos Farmacológicos Sc, Chihuahua City
  - Instituto Veracruzano en Investigación Clínica S.C., Veracruz
- Puerto Rico (2):
  - Advanced Clinical Research, LLC, Bayamón
  - GCM Medical Group, PSC - Hato Rey Site, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Effect of Retatrutide Compared With Semaglutide in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Metformin With or Without SGLT2 Inhibitor (TRANSCEND-T2D-2) — https://trials.lilly.com/en-US/trial/461538